CLINICAL TRIAL: NCT04897321
Title: B7-H3-Specific Chimeric Antigen Receptor Autologous T-Cell Therapy for Pediatric Patients With Solid Tumors (3CAR)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3CAR; NCI-2021-10933 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Solid Tumor; Osteosarcoma; Rhabdomyosarcoma; Neuroblastoma; Ewing Sarcoma; Wilms Tumor; Adrenocortical Cancer; Desmoplastic Small Round Cell Tumor; Germ Cell Cancer; Rhabdoid Tumor; Clear Cell Sarcoma; Hepatoblastoma; Melanoma; Carcinoma; Malignant Peripheral Nerve Sheath Tumors; Soft Tissue Sarcoma
MeSH Terms: conditions — Osteosarcoma; Rhabdomyosarcoma; Neuroblastoma; Sarcoma, Ewing; Wilms Tumor; Adrenal Cortex Neoplasms; Desmoplastic Small Round Cell Tumor; Neoplasms, Germ Cell and Embryonal; Rhabdoid Tumor; Sarcoma, Clear Cell; Hepatoblastoma; Melanoma; Carcinoma; Neurofibrosarcoma; Sarcoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Phase (Other): During the treatment phase, the participant receives an infusion of the B7-H3-CAR T cells that were made in the Collection and Manufacturing Phase. Chemotherapy is given for several days prior to the cellular infusion. Patients are then monitored for possible side effects, as well as effects of the treatment on their cancer.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: MESNA; Drug: B7-H3 CAR T cells

INTERVENTIONS:
Drug: Fludarabine — Fludarabine phosphate is a synthetic purine nucleoside analog. It acts by inhibiting DNA polymerase, ribonucleotide reductase and DNA primase by competing with the physiologic substrate, deoxyadenosine triphosphate, resulting in inhibition of DNA synthesis. Intravenous
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard derivative. It acts as an alkylating agent that causes cross-linking of DNA strands by binding with nucleic acids and other intracellular structures, thus interfering with the normal function of DNA. Intravenous
  Other Names: Cytoxan
Drug: MESNA — Mesna is a synthetic sulfhydryl (thiol) compound. Mesna contains free sulfhydryl groups that interact chemically with urotoxic metabolites of oxaza-phosphorine derivatives such as cyclophosphamide and ifosfamide
  Other Names: Mesnex
Drug: B7-H3 CAR T cells — The study participant will receive B7-H3-CAR T cells by vein, through either an IV or a central line.
  Other Names: CAR T- cell infusion

SUMMARY:
3CAR is being done to investigate an immunotherapy for patients with solid tumors. It is a Phase I clinical trial evaluating the use of autologous T cells genetically engineered to express B7-H3-CARs for patients ≤ 21 years old, with relapsed/refractory B7-H3+ solid tumors. This study will evaluate the safety and maximum tolerated dose of B7-H3-CAR T cells.The purpose of this study is to find the maximum (highest) dose of B7-H3-CAR T cells that are safe to give to patients with B7-H3-positive solid tumors.

Primary objective

To determine the safety of one intravenous infusion of autologous, B7-H3-CAR T cells in patients (≤ 21 years) with recurrent/refractory B7-H3+ solid tumors after lymphodepleting chemotherapy

Secondary objective

To evaluate the antitumor activity of B7-H3-CAR T cells

Exploratory objectives

* To evaluate the tumor environment after treatment with B7-H3-CAR T cells
* To assess the immunophenotype, clonal structure and endogenous repertoire of B7-H3-CAR T cells and unmodified T cells
* To characterize the cytokine profile in the peripheral blood after treatment with B7-H3-CAR T cells

DETAILED DESCRIPTION:
Treatment will include a single infusion of B7-H3-CAR T cells after lymphodepleting chemotherapy, with dosing based on the number of CAR+ T cells and patient weight. The study will evaluate the safety and maximum tolerated dose (MTD) of B7-H3-CAR T cells, using a standard 3+3 study design and a 6-week evaluation period. The total study duration will be 1 year, at which point patients will enroll on our existing institutional long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

Procurement and T-cell production eligibility*

*a previously collected, autologous leukapheresis product can be used for T-cell production

* Age ≤21 years old
* B7-H3+ solid tumor with measurable disease; B7-H3 expression will be evaluated by standard immunohistochemistry (IHC) using a previously obtained biopsy; a tumor is considered B7-H3 positive with an H-score ≥100
* Estimated life expectancy of >12 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥50
* For females of child bearing age:
* Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
* Not lactating with intent to breastfeed
* Meets eligibility criteria to undergo autologous apheresis, or have previously undergone autologous apheresis

Exclusion Criteria:

* Known primary immunodeficiency
* Known HIV positivity
* Severe intercurrent bacterial, viral or fungal infection (e.g. active hepatitis B or C infection or adenovirus infection)
* History of hypersensitivity reactions to murine protein-containing products
* Rapidly progressive disease (in the opinion of the study PIs)

Inclusion criteria

Treatment eligibility

* Age ≤21 years old
* B7-H3+ solid tumor with measurable disease
* Evidence of relapsed or refractory disease after standard first-line therapy
* Estimated life expectancy of >8 weeks
* Karnofsky or Lansky (age-dependent) performance score≥50
* Echocardiogram with a ventricular ejection fraction
* >40%; or shortening fraction ≥25%
* Adequate renal function defined as creatinine clearance or radioisotope GFR 50 ml/min/1.73m2 (GFR 40 ml/min/1.73m2 if < 2 years of age)
* Adequate pulmonary function defined as pulse oximetry ≥92% on room air or forced vital capacity (FVC) ≥50% of predicted value
* Total Bilirubin ≤3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤5 times the upper limit of normal for age
* Hemoglobin≥ 7g/dL (can be transfused)
* Platelet count >50,000/uL (can be transfused)
* Absolute neutrophil count (ANC) ≥ 1000/uL
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For females of child bearing age:
* Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
* Not lactating with intent to breastfeed
* If sexually active, agreement to use birth control until 3 months after T-cell infusion. Male partners should use a condom.
* Available autologous transduced T-cell product that has met GMP release criteria
* Agreement to participate in long-term follow-up protocol for patients, who have received genetically modified cell products

Exclusion criteria

* Known primary immunodeficiency
* History of HIV infection
* Severe, uncontrolled intercurrent bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products
* Receiving systemic steroid therapy exceeding the equivalent of 0.5 mg/kg/day of methylprednisolone, in the 7 days prior to B7-H3-CAR T-cell infusion
* Receiving systemic therapy in the 14 days prior to CAR T-cell infusion, which will interfere with the activity of the B7-H3-CAR product (in the opinion of the study PIs).
* Rapidly progressing disease (in the opinion of the study PIs)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety of B7-H3-CAR T cells | 6 weeks after B7-H3-CAR T cell infusion
  A phase I design to determine the maximum tolerated dose (MTD) of autologous, B7-H3-CAR T cells. Four dose levels (3x10^5/kg, 1x10^6/kg, 3x10^6/kg, and 1x10^7/kg) will be evaluated.

SECONDARY OUTCOMES:
Clinical Response | 6 weeks after B7-H3-CAR T cell infusion
  The number of patients with objective responses (complete response (CR) + partial response (PR)) determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Chris DeRenzo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols